CLINICAL TRIAL: NCT04961177
Title: Increasing Use of Earned Income Tax Credit (EITC) in New Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Janet M Page-Reeves, Associate Professor, University of New Mexico
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 21-123
Record Dates: First submitted 2021-06-22; First posted 2021-07-14 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Adverse Childhood Experiences
Keywords: EITC; Poverty; ACEs; Frontline Health Workers; Community Health Workers (CHWs)
MeSH Terms: interventions — Mass Screening; Insemination, Artificial, Heterologous

STUDY DESIGN:
Intervention Model Description: The proposed intervention will have five components:
  1. We will conduct trainings for our partner agencies and their frontline health workers to increase knowledge and understanding of: 1.) Risk/protective factors for ACEs and 2.) Eligibility criteria and filing requirements and procedures for EITC.
  2. Working with our partners, we will also conduct EITC educational outreach and information sessions targeted to potential EITC filers.
  3. We will track program level EITC data regarding screening and assistance provided to clients by CHWs in our network and the number of clients who submit EITC claims and the amounts received.
  4. We will conduct a pre/post survey with clients who submit EITC claims to determine whether EITC reduces risk factors and increases protective factors for ACEs.
  5. We will disseminate this model throughout the state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EITC & ACEs Training (Other): Trainings for frontline health workers about EITC and ACEs.
  Interventions: Other: EITC & ACEs Training
- EITC Outreach and Screening (Other): Our partners will implement EITC outreach events and EITC screening with clients.
  Interventions: Other: EITC Outreach & Screening
- EITC Assistance (Other): Our partners will screen clients for EITC and refer those who qualify for free tax preparation assistance and assistance submitting their tax returns.
  Interventions: Other: Assistance with EITC

INTERVENTIONS:
Other: EITC & ACEs Training — We will deliver up to 56 trainings to 65 frontline health workers and 25 staff of our partner organizations. The training will include: 1.) Information about what ACEs are, and the risk and protective factors associated with ACEs and 2.) Information regarding EITC benefits, eligibility, application procedure and logistics, referrals for free tax preparation assistance, and use of EITC tools., and 3.) frontline health workers will receive additional training in protocols for reporting to support Objective #2.
  Arms: EITC & ACEs Training
Other: EITC Outreach & Screening — Our partners will screen and refer a minimum of 5200 clients (65 CHWs x 10 clients per quarter x 2 years) for EITC. Our evaluation team will track the number of individuals screened, the number found to be eligible/not eligible, the number referred out and to which free tax prep service, and if available, the number who use the free tax prep service, the number who file a tax claim for EITC, the number who receive EITC benefits, and the amount of the benefit.
  We will conduct community-level EIT outreach by integrating EITC outreach and education into planned community events in the neighborhoods and service areas of our partners. The events will provide information about the EITC to the public. We will have a minimum of 48 events to reach a minimum of 480 potential filers (48 events x 10 participants each).
  Arms: EITC Outreach and Screening
Other: Assistance with EITC — We will conduct a statistical analysis of the impact of EITC funds on ACEs risk and protective factors in the lives of EITC benefit recipients. Project CHW team members will invite 200 clients who qualify to receive EITC benefits to participate in the study using an approved recruitment script. With those who agree to participate, the CHW team member will obtain consent and administer a baseline survey. A post-survey will be administered at 4 months.
  In addition, we will gather qualitative data to help us understand impacts of this project. The post-survey will contain an open/qualitative response question asking participants to describe how the EITC benefit impacted them, how they felt when they received it, how important it was, and what they did with the funds. In Y2, the Research Team will conduct interviews with a subset of 20 clients who participated in the pre/post survey.
  Arms: EITC Assistance

SUMMARY:
Purpose of the Proposed Project. The literature makes clear that poverty and financial hardship and lack of social support are significant risk factors that create a household environment conducive to Adverse Childhood Experiences (ACEs). The purpose of the project is to reduce ACEs-related risk factors that threaten child wellbeing in the homes of low-income families by maximizing Earned Income Tax Credit (EITC) claims among populations of focus in Bernalillo County, and disseminating successful strategies for risk-reduction throughout the state. The project team will do this by integrating outreach and education regarding ACEs and EITC benefits across a group of community-based initiatives, training programs, networks, and collaborators that work with frontline health workers [Community Health Workers (CHWs) and Medical Assistants (MAs)].

DETAILED DESCRIPTION:
Goal. The goal of this project is to reduce risk factors and increase protective factors for ACEs by measurably reducing household financial strain, financial insecurity, and economic instability, and increasing social support for low-income populations of focus in Bernalillo County (with an emphasis on designated Economic Opportunity Zones (EOZs) as required by the award) by increasing EITC utilization. The team will accomplish this using an innovative strategy to mobilize frontline health workers to conduct EITC outreach, education, referral, and support across our robust community-based initiatives, collaborations, networks, and training programs, and to disseminate this model for increasing EITC utilization.

Objectives. This project has three objectives.

1. Objective 1. By Y1, M12, increase capacity for EITC outreach and education among 28 core, established, multi-sectoral partner agencies by engaging them in the planning, design, and implementation to 56 trainings for frontline health workers and staff as measured by: A.) Improvement in scores on a pre/post test administered to 65 frontline health workers and 25 partner agency staff before and after the training regarding knowledge and understanding of ACEs-related risk and protective factors and EITC benefits, eligibility, logistics, and referral. B.) Documented increase in the number of times agency frontline health workers and staff use existing EITC materials from national EITC campaigns or the Internal Revenue Service website or start to use the tools following the training.
2. Objective 2. By Y3, M6, increase EITC utilization in Bernalillo County by a minimum of 5200 new EITC filed claims during the project implementation period by tax filers who have not previously filed for EITC in the past 12 months by mobilizing our partners and their 65 CHWs to conduct EITC education, outreach, screening and referral for free tax preparation assistance (65 CHWs x 10 clients per quarter x 2 years), and co-sponsorship of a minimum of 48 community outreach events reaching a minimum of 480 potential EITC filers (48 events x 10 filers).
3. Objective 3. By Y3, M12, using a rigorous evaluation of project activities and outcomes, demonstrate a statistically significant change in ACEs risk/protective factors between baseline and four months among a cohort of 200 EITC filers in order to demonstrate evidence that mobilizing community agencies and frontline health workers is a strong model for increasing EITC utilization: A.) Demonstrate a decrease in household financial strain, financial insecurity, and household economic instability as measured by a change in mean score of at least 0.77 on the In Charge Financial Distress/Financial Well-being Scale (IFDFW). B.) Demonstrate an increase in informational social support as measured by the informational support questions from the Medical Outcomes Study Social Support Survey (MOS-SSS).

Outcome and Impact. The outcome of this project will be to create a cadre of trained frontline health workers and community agencies with the knowledge and capacity to provide EITC outreach, information, screening, and referrals to low-income clients to increase utilization of EITC in New Mexico. The anticipated impact of this effort will be that more New Mexicans will file EITC claims and the funds they receive will help to ameliorate the stress of financial hardship and reduce poverty. Furthermore, the experience of working with the frontline health worker will increase social support and utilization of EITC, both of which will reduce negative social determinants of health and risk factors for ACEs and increase preventive factors for ACEs of children who live in some of the most at-risk homes, improving the wellbeing of these children today and creating a foundation for them to have healthier lives as adults.

ELIGIBILITY:
Inclusion Criteria

* Adult, 18 or over
* Speak English or Spanish
* Work as a frontline health worker or staff at one of our partner agencies who takes our training
* Be a client of one of the frontline health workers of our partner agencies who qualifies for EITC who has not submitted an EITC claim in the past 12 months and is interested in receiving assistance to submit an EITC claim through our project

Exclusion Criteria

* Children --individuals younger than 18
* Fetuses
* Individuals unable to provide consent
* Individuals who are incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
A: Financial strain and insecurity. | 4 months
  We will measure change in financial strain, financial insecurity, and economic instability among clients who are at high risk for Adverse Childhood Experiences (ACEs) and who submit an EITC claim as a result of assistance from this project. Financial strain, financial insecurity, and economic instability will be measured as demonstrated by a minimum of a 0.77 point change on the In Charge Financial Distress/Financial Well-being Scale (IFDFW), with an expected change of 1.5 - 2 points.
B: Informational Social Support | 4 months
  We will measure change in informational support that occurs as a result of frontline health workers providing outreach, education, and screening for EITC, and referral for free tax help. We will measure change in informational support using the MOS-SSS Informational Support subscale. We hypothesize a minimum change of 1.5 points.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Page-Reeves, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT04961177/ICF_000.pdf